CLINICAL TRIAL: NCT05946018
Title: Physiatrist Ergonomic Intervention on Work Related Musculoskeletal Pain in Surgeons: A Randomized Control Trial
Brief Title: Physiatrist Ergonomic Intervention on Work Related Musculoskeletal Pain in Surgeons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Kimberly Kho, MD, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU-2023-0516
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Musculoskeletal Pain; Work Related Stress; Quality of Life; Grip
MeSH Terms: conditions — Musculoskeletal Pain; Occupational Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Education only (Other): This arm only includes a 6-8 minute educational video on ergonomics.
  Interventions: Other: Educational video on ergonomics
- Education and coaching sessions (Other): This arm includes a 6-8 minute education video on ergonomics and 1:1 15 minute coach sessions at 0, 2, 4, and 6 weeks.
  Interventions: Other: Educational video on ergonomics; Other: Verbal physical therapy coaching sessions

INTERVENTIONS:
Other: Educational video on ergonomics — A 6-8 minute education video that includes information on why ergonomics is important and recommendations for how to arrange the operating room to reduce the risk of injury.
Other: Verbal physical therapy coaching sessions — Physical therapy coaching sessions include a standard assessment with individualized instruction on range of motion, strength, endurance, and flexibility.
  Arms: Education and coaching sessions

SUMMARY:
The goal of this randomized control trial is to learn if physical therapy coaching and education improves work-related muscle pain in surgeons more than education alone. The main focuses of this study are to:

1. To evaluate pain in surgeons before and after surgical cases.
2. To evaluate work-load related stress in surgeons after surgical cases.
3. To evaluate surgeons' quality of life.
4. To evaluate surgeons' grip strength.

Participants will be put into two groups at random. One group will watch an educational video only. The other group will watch an educational video and get a coaching session from a physical therapist.

DETAILED DESCRIPTION:
All participants will undergo the same baseline, pre-intervention assessments. Pre-intervention assessments will include several questionnaires: general demographic questionnaire, baseline questionnaire, WHO GPAQ for assessment of physical activity, and AROM assessment. Additionally, following one day operating they will complete a SURG-TLX questionnaire, Brief Pain Index (BPI), and a questionnaire regarding how many hours they operated that day and what type of surgeries they performed (Surgery Day Questionnaire).

For participants randomized to the education only group, they will watch a short (5-7 minute) educational video. The video content includes information on why ergonomics is important (preventing work-related musculoskeletal disorders, types of injuries, physician longevity) and recommendations for how to ergonomically arrange the operating room to reduce the risk of injury.

For participants randomized to the education plus personal coaching group, they will first watch the same video as described previously. Then they will have four 15 to 20-minute sessions with a physiatrist. These sessions will include a standard assessment with individualized instruction on range of motion, strength, endurance, and flexibility. These sessions will include verbal coaching, instructor demonstration, however no hands-on treatment or intervention will be provided. The sessions will occur at 0 weeks (same day as participant views video), 2 weeks, 4 weeks, and 6 weeks after viewing of the educational video. The first session will be in person, the remainder of the sessions will be virtual.

Post-intervention follow up will begin after the video is viewed by those in the education-only group and after the video is viewed and the first personal coaching session is complete by the education plus coaching group. The first timepoint of post-intervention assessment will be the first operating day after the intervention. Assessments will include SURG-TLX, BPI, and Surgery Day Questionnaire. Two additional post-intervention assessments will be at 2 weeks after initial intervention and 6 weeks after initial intervention. The 6 week timepoint reflects the completion of the personal coaching series for those in that group.

Long-term follow-up assessments will be performed at 3 and 6 months after the initial intervention (week 0). The assessments that will be administered then will include a demographic/general questionnaire, WHO GPAQ, SURG-TLX, BPI, and Surgery Day Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Attending/faculty surgeon or surgical trainee (PGY2 or above) in any surgical specialty
* Operates at least one day per week

Exclusion Criteria:

* Currently under active treatment for a musculoskeletal injury (example: physical therapy)
* Plans to decrease operating time to less than one day per week in the next 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
To evaluate pain in surgeons after operating. | 6 months
  Surgeons receiving personalized education and a physical activity plan will report less pain (as assessed by the Brief Pain Index). The BPI measures pain on a 0-10 scale with higher scores meaning worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Kho, MD, Principal Investigator — UTSW
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No